CLINICAL TRIAL: NCT01402635
Title: A Randomized Controlled Trial Comparing Central Laboratory and Point-of-care Chemistry Test for Solving the Emergency Department Crowding
Brief Title: Can the Point-Of-Care Chemistry Test (POCT) Solve the Emergency Department (ED) Crowding?
Acronym: POCTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Do Shin, Associated professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SNUEMS201101
Record Dates: First submitted 2011-01-09; First posted 2011-07-26 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Crowding
Keywords: crowding; Point-of-Care Systems; emergency medicine
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- POCT lab (Experimental): The patient group whose laboratory test perform by POCT chemistry analyzer.
  Interventions: Device: point-of-care chemistry test(POCT) (Piccolo)
- central laboratory group(CLT) (Active Comparator): The patients group whose laboratory test perform by central laboratory.
  Interventions: Device: point-of-care chemistry test(POCT) (Piccolo)

INTERVENTIONS:
Device: point-of-care chemistry test(POCT) (Piccolo) — comprehensive chemistry POCT including ALB, ALP, ALT, AST, BUN, Ca, Cl-, Cre, Glu, K+, Na+, TBil, TCO2, TP It takes 12minutes to perform analyze.
  Other Names: Piccolo® xpress; Piccolo® Comprehensive Metabolic Reagent Disc

SUMMARY:
The hypothesis of this study that the Point-Of-Care Chemistry Test (POCT) may shorten Emergency Department (ED) length of stay (LOS).

DETAILED DESCRIPTION:
ED crowding is one of the most serious problems in ED. POCT has shorter turn-around time compared to centralized laboratory system. If POCT introduce to ED, it may help to shorten LOS of ED patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years
* clinically required to have chemistry lab tests
* ESI 2-5
* written agreement to participate

Exclusion Criteria:

* no agreement
* ESI level 1
* no chemistry lab

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10244 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
length of stay | average 7days from ED visit(up to time of discharge at ED or admission to ward)
  Time interval between registration at ED and leaving at ED(discharge, admission, etc.)

SECONDARY OUTCOMES:
length of stay(subgroup) | average 7days from ED visit (up to time of discharge at ED or admission to ward)
  length of stay analysis for Emergency Severity Index (ESI) 3-4, admission or discharge group

CONTACTS AND LOCATIONS:
Overall Officials: Sang Do Shin, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Lee EJ, Shin SD, Song KJ, Kim SC, Cho JS, Lee SC, Park JO, Cha WC. A point-of-care chemistry test for reduction of turnaround and clinical decision time. Am J Emerg Med. 2011 Jun;29(5):489-95. doi: 10.1016/j.ajem.2009.11.020. Epub 2010 Apr 24. PMID 20825817